CLINICAL TRIAL: NCT01418391
Title: the Effect of the Transversus Abdominis Plane (TAP) Block on the Minimal Laparotomy : a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Hung-Te Hsu/ Department of Anesthesia, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KMUH-IRB-990400; KMUH-IRB-990400 (Other: KaohsiungMU)
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-05

CONDITIONS: Colon Cancer
Keywords: minimal laparotomy; TAP block; morphine consumption; post-operative analgesia
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- morphine consumption (Experimental)
  Interventions: Procedure: Transversus Abdominis Plane block

INTERVENTIONS:
Procedure: Transversus Abdominis Plane block — TAP BLOCK:
  dosage form: 0.5% bupivacaine 75mg with 2% xylocaine 300 mg mixed dosage: total 30 ml frequency: single shot duration: 12~18 hours upon to the regional anesthetics choose
  Other Names: TAP block

SUMMARY:
Transversus abdominis plane block (TAP block) is a new regional block for abdominal wall.It had been reported the effect of post-operative pain control in minor abdominal surgery, such as inguinal hernia repair and appendectomy. On the other hand, because of the accurate of the pre-operative images, the minimal laparotomy for colon cancer was accomplished. Thus, the purpose of this study is to investigate the effect, such as analgesic effect, hemodynamic stability, and post-operative morphine consumption, of TAP block in minimal laparotomy.

DETAILED DESCRIPTION:
outcome measures:

* Hemodynamic parameters (mean artery pressure, heart rate): recorded at time points of before induction of general anesthesia (baseline), after tracheal intubation immediately, after surgery started 1, 2, 3, 4, 5, 10, 15, 20, 25, and 30 min; then recorded them every 10 mins.
* Post-operative morphine consumption: recorded morphine consumption at the time intervals of post-operative 0~6 h, 6~12 h, 12~24 h, 24~36 h, and 36~48 h ,respectively. The total amount of morphine consumption was also counted.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists physical status I-III, ≧ 18 years of age, and needed double-lumen endotracheal tube (DLT) for thoracic surger

Exclusion Criteria:

* increased risk for regurgitation and pulmonary aspiration, history of gastroesophageal reflux, and pregnancy
* a tracheostomy or prolonged ventilation on ICU was planned, patients were also excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
amount of post-operative morphine consumption | post-operative 48 hours

SECONDARY OUTCOMES:
evaluation of post-operative pain status using visual analog scale (VAS) and superimposed face pain severity scale | post-operative 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Te Hsu, VS, Principal Investigator — Department of anesthesia, Kaoshiung medical university hospital
Locations (1):
- department of anesthesia, Kaohsiung medical university memorial hospital, Kaohsiung City, Kaohsiung, Taiwan